CLINICAL TRIAL: NCT07272694
Title: A Prospective Controlled Clinical Study Evaluating the Effect of Bone and Autologous Dentin Grafting in the Osteotomy Gap During the Split Crest Procedure With Simultaneous Implant Placement
Brief Title: Split Crest Procedure: Is It Necessary to Fill the Gap?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vladimir Biocanin (Other)
Responsible Party: Sponsor-Investigator, Vladimir Biocanin, Principal Investigator, Faculty of Stomatology in Pancevo
Organization: Faculty of Stomatology in Pancevo (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SC-DENTIN-2024-01
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Alveolar Bone Resorption; Alveolar Bone Grafting; Bone Expansion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Split Crest Only (Active Comparator)
  Interventions: Procedure: Split Crest Technique
- Split Crest + Bone Graft (Experimental)
  Interventions: Procedure: Split Crest Technique
- Split Crest + Dentin Graft (Experimental)
  Interventions: Procedure: Split Crest Technique

INTERVENTIONS:
Procedure: Split Crest Technique — A surgical split crest (alveolar ridge splitting) procedure performed to increase horizontal alveolar bone width and enable simultaneous dental implant placement. A controlled osteotomy is created along the crest of the ridge, followed by gradual expansion of the buccal cortical plate to form an osteotomy gap for implant insertion.

SUMMARY:
This prospective controlled clinical study evaluates the effectiveness of adding bone graft or dentin graft material during the split crest (alveolar ridge splitting) procedure for horizontal ridge augmentation with simultaneous implant placement.

The study includes patients with narrow alveolar ridges requiring implant-supported rehabilitation. Participants are divided into three groups: split crest without grafting, split crest with bone graft, and split crest with dentin graft. The aim is to determine whether the addition of graft material to the osteotomy gap improves bone width, bone density, and primary implant stability compared to the split crest technique alone.

Clinical and radiographic assessments are performed using cone-beam computed tomography (CBCT) and implant stability measurements (ISQ values) before surgery, immediately after implant placement, and three months postoperatively. All patients are monitored over a one-year follow-up period to evaluate healing progression and treatment outcomes.

This study seeks to identify the most effective approach for horizontal ridge augmentation and to improve clinical decision-making in implant dentistry. The findings aim to contribute to optimizing surgical protocols, enhancing implant stability, and improving long-term functional outcomes for patients.

Participation is voluntary, and all procedures are conducted in accordance with approved ethical standards and clinical guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-65 years
* Indication for tooth extraction in posterior mandibular region with planned implant placement
* Presence of post-extraction alveolar bone defect requiring ridge preservation procedure
* Good general health (ASA I or ASA II)
* Ability to understand the study procedures and provide written informed consent
* Willingness to comply with scheduled follow-up visits and study protocol

Exclusion Criteria:

* Systemic diseases affecting bone healing (e.g. uncontrolled diabetes, osteoporosis, metabolic bone disorders)
* History of radiotherapy in the head and neck region
* Use of bisphosphonates or other antiresorptive medications
* Active periodontal or periapical infection at the surgical site
* Heavy smokers (>10 cigarettes per day)
* Pregnancy or breastfeeding
* Known allergies to materials used in the study
* Poor oral hygiene or lack of complianc

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Change in alveolar ridge width following split crest proceduree with or without bone or dentin grafting | Preoparative, Immediately postoperative, and 3 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Stomatology, Department of Oral Surgery, University Business Academy in Novi Sad,, Pančevo, Serbia

IPD SHARING:
Plan to Share IPD: No